CLINICAL TRIAL: NCT04681209
Title: Increasing Children's Defending Behaviors: Using Deviance Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Wendy P. Gordon, Principle Investigator, Auburn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: AuburnUDRT
Record Dates: First submitted 2020-12-14; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Bullying of Child
Keywords: Peer Relationship; Bullying Prevention

STUDY DESIGN:
Intervention Model Description: Schools were randomly assigned to have their fourth-grade and fifth-grade classrooms participate in either a DRT-based intervention activity or a traditional (i.e., empathy-based) intervention activity.
Who Masked: Participant, Outcomes Assessor
Masking Description: Schools (including teachers and students) were not aware of whether they were receiving an experimental or traditional intervention activity. Those collecting the data were also not aware of the experimental condition of the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DRT-Condition (Experimental): This is the experimental group that engaged in the DRT-based intervention activity.
  Interventions: Behavioral: DRT Condition
- Empathy-Condition (Active Comparator): This is the experimental group that engaged in the empathy-based intervention activity.
  Interventions: Behavioral: Empathy Condition

INTERVENTIONS:
Behavioral: DRT Condition — Children were asked to provide five descriptors of two children who each engaged in defending behaviors. Two weeks later they were told the top seven descriptors given by the hundreds of children participating in the project. This was followed by a brief discussion of how one could best help another kid who was getting bullied. Children then made posters to share with younger grades as to what "friendship heroes" are like, using the descriptor words shared with them, and how to be a friendship hero (i.e., how to help someone who is being bullied). Posters were hung for two-to-four months after the intervention activity.
  Arms: DRT-Condition
Behavioral: Empathy Condition — Children in the empathy-based condition were asked to provide five descriptors of how two children who were bullied would fee. Two weeks later they were told the top seven descriptors given by the hundreds of children participating in the project. This was followed by a brief discussion of how one could best help another kid who was getting bullied. Children then made posters to share with younger grades as to what being bullied feels like, using the descriptor words shared with them, and how to be a friendship hero (i.e., how to help someone who is being bullied). Posters were hung for two-to-four months after the intervention activity.
  Arms: Empathy-Condition

SUMMARY:
The National Institute of Child Health and Human Development (NICHD) has identified bullying as a significant public health concern. The research tests a novel approach to increase children's defending of victims of bullying. Previous research has shown that the presence of defenders leads to decreases in bullying. Thus, promoting defending has become a critical component of anti-bullying interventions. However, how to best motivate defending has been relatively unstudied. Deviance Regulation Theory (DRT) provides a theoretical basis for motivating positive health and social behaviors. This theory proposes that individuals are motivated to behave in ways that differentiate them from others in a positive manner. Accordingly, individuals will be motivated to engage in a behavior if they believe the behavior occurs infrequently and will be viewed positively by others. As children report that few of their peers defend victims of bullying, the goal of this study is to increase defending by communicating to children that defenders possess traits valued by their peers (e.g., being popular, kind). Children in 4th-grade and 5th-grade classrooms received a DRT-based anti-bullying intervention or an anti-bullying intervention focused on increasing empathy for victims and strategies for defending peers. Data collection occurred three times during the school year: a) at baseline, two weeks prior to the intervention; b) 3 months post-intervention; and c) 6 months post-intervention. Findings showed that compared to the traditional anti-bullying intervention, the DRT-based intervention resulted in larger, more sustained gains in teacher-reported defending, but not peer-reported or self-reported defending. Contrary to expectations, gains in teacher-reported defending were greatest for children who viewed defending to be normative amongst their classmates. Increases in defending were also greatest among those children least likely to defend (i.e., those low in popularity and prosocial behavior, and those often bullied by peer). These findings have implications for the development of anti-bullying interventions and more broadly for understanding how to encourage important behavioral changes in childhood and adolescence. However, more research is needed to understand why increases were limited to only defending behaviors observable to teachers.

DETAILED DESCRIPTION:
This study, conducted over the 2017-2018 and 2018-2019 school years examined whether a DRT-based intervention activity resulted in greater increases in defending behaviors in response to witnessed bullying than a more traditional, empathy-based activity. Thirteen schools were randomly assigned to receive either the DRT-based or empathy-based activity, and all fourth-grade and fifth-grade children were invited to participate. Defending behaviors were assessed approximately two weeks prior to participation in the activity and at three-month and six-month follow-ups. Data collected included peer-reports, teacher-reports, and self-reports. Also examined was whether popularity, peer acceptance, prosocial behavior, peer victimization, empathy, self-efficacy for defending, moral disengagement, or gender moderated intervention effects.

ELIGIBILITY:
Inclusion Criteria:

* Child in the fourth-grade or fifth-grade of participating schools

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1564 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Changes in Peer-reported Defending across The School Year | three-month follow-up; six-month follow-up
  Peer ratings of how often each participating classmate defended bullied peers
Changes in Self-reported Defending across the School Year | three-month follow-up; six-month follow-up
  Children's ratings of how often they defended bullied peers
Changes in Teacher-reported Defending across the School Year | three-month follow-up; six-month follow-up
  Teachers' ratings of how often each participating student defended bullied peers

SECONDARY OUTCOMES:
Changes in Perceptions of Defenders across The School Year | three-month follow-up; six-month follow-up
  Children's ratings of how much children who help others who are bullied are popular, kind, sensitive to other's feelings, leaders, well-liked, confident, and helpful. Higher scores reflected more positive perceptions of children who defend.
Changes in Peer Aggression across the School Year | three-month follow-up; six-month follow-up
  Ratings participating children received from classmates on the items "calls other kids bad names or say mean things to them," "tell other kids they can't play with them or won't be friends with them," and "hit or push other kids." Ratings were made on a scale from never to a lot. Ratings received from participating classmates were averaged, and item scores were averaged to compute a composite aggression score with higher scores indicating higher levels of aggressive behavior.
Changes in Peer Victimization across the School Year | three-month follow-up; six-month follow-up
  Ratings received from participating classmates on the items "get left out of things that kids are doing (kids don't let him or her play with them), "get hit or pushed," and "kids call [this child] bad names or say mean things to him or her." Items were rated on a scale from never to a lot. Ratings received from all participating classmates are averaged for each item, and item scores are averaged to create a composite peer victimization score. Higher scores indicated higher levels of peer victimization.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy P Gordon, Principal Investigator — Auburn University
Locations (1):
- Auburn University, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Only de-identified data from all 1,564 participants will be shared

REFERENCES:
- [Result] Troop-Gordon W, Frosch CA, Wienke Totura CM, Bailey AN, Jackson JD, Dvorak RD. Predicting the development of pro-bullying bystander behavior: A short-term longitudinal analysis. J Sch Psychol. 2019 Dec;77:77-89. doi: 10.1016/j.jsp.2019.10.004. Epub 2019 Nov 25. PMID 31837730